CLINICAL TRIAL: NCT05673616
Title: MRI-Based Structural Changes in Lumber Spine in Subjects With Discogenic Low Back Pain After Mckenzie Exercises.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FUI/CTR/2022/3
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Mechanical Low Back Pain
Keywords: Physical therapy; Intervertebral disc; Magnetic resonance imaging; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Inclusion Criteria
  1. Patients having Discogenic LBP referred from hospital.
  2. Male and female both
  3. Ptients hving Modic changes in MRI.
  3.Otherwise, healthy patients with age range from 18 to 55 years.
  Exclusion criteria:
  1. Patients with non-mechanical LBP
  2. Patients not meeting age range
  3. Patients with any major co-morbidity
  4. Any type of systemic illness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Mckenzie Extension Exercises
  Interventions: Other: Mckenzie Extension Exercises

INTERVENTIONS:
Other: Mckenzie Extension Exercises — After two weeks of initial consultation, the patient will be taught to perform slouch-overcorrect on day 1 followed by flexion on day 2 in lying position and accompanied by flexion for 5 days in sitting position and finally flexion in standing will be performed.
  The exercises will be repeated for 10 times and followed by extension in standing exercises.

SUMMARY:
In the rehabilitation department, we are working with patients of low back pain for routine management and as well as for research. Still now, the biomechanical ground proofing the beneficial effects of McKenzie Mechanical diagnosis and therapy on non-mechanical low back pain has not been studied in depth. This qausi-experimental study will provide expert-level evidence using gold standard MRI findings to add McKenzie MDT in routine treatment of the condition.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study will be:

1. To determine the effects of McKenzie Mechanical Diagnosis and Therapy (MDT) on MRI-based structural changes in Pateints with mechanical low back pain.
2. To determine the effects of McKenzie MDT on Pain and Disabaility scores in patients with mechanical low back pain.
3. To determine the effects of McKenzie MDT on Disabaility scores in patients with mechanical low back pain.

HYPOTHESIS:

Alternate Hypothesis:

The Mckenzie MDT will be effective in improving the MRI-based structural changes, pain and disability caused by the mechanical low back pain.

Null Hypothesis:

The Mckenzie MDT will not be effective in improving the MRI-based structural changes, pain and disability caused by the mechanical low back pain.

Research Design: Quasi - experimental Study.

Clinical setting: Foundation University College of Physical Therapy, Foundation University Islamabad.

Study duration: 12 months

Sampling technique: Non-probability Purposive sampling

Intervention to be given

After assessing the patient for eligibility, following intervention regime will be followed:

1. st consultation-Day 1: In standing right side gliding will be repeated for ten to twenty times. Afterwards, extension will be repeated in lying position for ten to twenty times.

   The protocol will be repeated after every three hours.
2. nd consultation- Day 3: Extension will be repeated in lying position for ten to twenty times. The protocol will be repeated after every three hours.
3. rd consultation- Day 15: After two weeks of initial consultation, the patient will be taught to perform slouch-overcorrect on day 1 followed by flexion on day 2 in lying position and accompanied by flexion for 5 days in sitting position and finally flexion in standing will be performed.

The exercises will be repeated for 10 times and followed by extension in standing exercises.

Significance:

McKenzie mechanical diagnosis and therapy (MDT) is more effective than other therapeutic physiotherapies. But, the biomechanical ground proofing of the beneficial effects of MDT on non-mechanical low back pain has not been studied in depth. This gap will be filled by the gold standard MRI imaging technology that allows non-invasive and more detailed view of intervertebral disc. This study will emphasize the healthcare practitioners regarding the cellular level benefits of said intervention and hence decrease the surgical cost by early treatment through physical therapy and rehabilitation.

This study will emphasize the healthcare practitioners regarding the cellular level benefits of said intervention and hence decrease the surgical cost by early treatment through physical therapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Both genders having low back pain. Patients having modic changes in MRI. Otherwise healthy patients with age range from 18 - 55 years.

Exclusion Criteria:

Patients with non-mechanical LBP Patients not meeting age range Patients with any major co-morbidity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
MRI changes | At baseline and 4 weeks
  fatty infiltration and modic changes

SECONDARY OUTCOMES:
Pain intensity assessed by numeric pain rating scale | At baseline and 4 weeks
  Pain will be assessed by numeric pain rating scale
Disability will be assessed by Roland-Morris Low Back Pain and Disability Questionnaire (RMQ) | At baseline and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan